CLINICAL TRIAL: NCT04189835
Title: EVITA Study - Epstein-Barr Virus Infection moniToring in renAl Transplant Recipients - Early Identification of Increased Risk of Infection and Cancer for Individualised Immunosuppression.
Brief Title: EVITA Study - Epstein-Barr Virus Infection moniToring in renAl Transplant Recipients
Acronym: EVITA
Status: Completed | Type: Observational
Sponsor: University of Aarhus (Other)
Collaborators: Rikshospitalet University Hospital (Other); Aarhus University Hospital (Other); Odense University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: EBV Renal
Record Dates: First submitted 2019-11-25; First posted 2019-12-06 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: EBV Infection; EBV Viremia; Epstein-Barr Virus Associated Lymphoproliferative Disorder; Post-transplant Lymphoproliferative Disorder
MeSH Terms: conditions — Epstein-Barr Virus Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma, whole blood and tissue biopsies.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Kidney transplant recipients: Adults and children undergoing kidney transplantation in Norway and the western part of Denmark.
  Interventions: Diagnostic Test: EBV DNA in whole blood and plasma

INTERVENTIONS:
Diagnostic Test: EBV DNA in whole blood and plasma — Consecutive measurements of EBV DNA in whole blood and plasma

SUMMARY:
Transplant recipients are treated with immunosuppressive drugs to avoid rejection of the transplanted organ. As the medication impairs the immune response, it also increases the risk of serious infections and cancer in transplant recipients compared with the general population.

Previous studies have shown a close association between Epstein-Barr virus (EBV) and post transplant lymphoproliferative disorder (PTLD), with frequent demonstration of the virus in lesional tissues. Transplant recipients without evidence of EBV infection prior to transplantation (EBV seronegative) are at particularly high risk of developing PTLD. Other risk factors include a high viral load. As part of a preventive approach against PTLD, several transplantation units now monitor the occurrence of EBV DNAemia after transplantation. However, there is little evidence to guide this strategy; nor is there consensus concerning either the best specimen to use for EBV analysis (whole blood or plasma) or the appropriate clinical action to take if EBV DNAemia is detected.

Our aim is to estimate the incidence and clinical consequences of Epstein-Barr virus (EBV) DNAemia in whole blood and plasma in renal transplant recipients, and to determine if persistence of EBV DNAemia can predict excessive immunosuppression as indicated by the incidence of infections requiring hospitalisation, EBV driven PTLD and mortality.

ELIGIBILITY:
Inclusion Criteria:

* Children from 2 years of age receiving a kidney transplant from a living or deceased donor.
* Adults 18 years or older who receive a kidney transplant from a living or deceased donor.
* Capable of giving written informed consent to participation in the study (legal guardians capable of giving written informed consent to participation in the study in case of children younger than 18 years old).

Exclusion Criteria:

* Patients unable to comply with the study requirements.
* Withdrawal of consent.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with end-stage renal disease in the southern part of Norway and in the western part of Denmark qualified to undergo kidney transplantation.
Sampling Method: Non-Probability Sample
Enrollment: 509 (Actual)
Dates: Start 2020-01-03 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
The incidence rate of EBV driven PTLD | 2 years
  The incidence rate of EBV driven PTLD in patients with 2 consecutive positive PCR samples for EBV DNA in whole blood and/or plasma during follow up (persistent EBV DNAemia). The detection level for EBV DNA in the whole blood is 110 IU/ml. Levels of EBV DNA < 1000 IU/ml are not quantified. The lower limit of detection for the EBV DNA plasma analysis is 25 IU/ml. Levels of EBV < 100 IU/ml are not quantified
The incidence rate of infections requiring hospitalisation in patients with persistant EBV DNAemia | 2 years
  The incidence rate of infections requiring hospitalisation in patients with 2 consecutive positive PCR samples for EBV DNA in whole blood and/or plasma during follow up (persistent EBV DNAemia).
Mortality rate in patients with persistant EBV DNAemia | 2 years
  Mortality rate in patients with 2 consecutive positive PCR samples for EBV DNA in whole blood and/or plasma during follow up (persistent EBV DNAemia).

SECONDARY OUTCOMES:
The incidence of symptomatic opportunistic infections | 2 years
  Defined as CMV, BK virus, Herpes simplex virus 1 and 2, Human herpes virus 6 and 7, and Varicella zoster virus. In addition, bacterial pathogens such as Legionella pneumophila, Listeria monocytogenes, Mycobacterium tuberculosis, Nocardia, all parasitic infections i.e. Pneumocystis jirovecii and fungal infections are regarded as opportunistic infections.
Incidence of infections requiring hospitalisation | 2 years
Incidence of EBV driven PTLD during follow-up. | 2 years
  PTLD verified by a biopsy. Cases of PTLD will be reviewed according to the WHO-definitions
Incidence of acute rejection | 2 years
  The incidence of acute rejection and chronic graft changes will be evaluated according to the Banff classification system. Cases without a biopsy will be registered if they have been treated as a an acute rejection
Kidney graft function | 2 years
  Kidney graft function at 2, 6, 12 and 24 months after transplantation will be evaluated by estimated glomerular filtration rate (eGFR, mL/min.) and urine albumin/creatinine

CONTACTS AND LOCATIONS:
Overall Officials: Bente Jespersen, Professor, Principal Investigator — Aarhus University Hospital
Locations (3):
- Denmark (2):
  - Aarhus University Hospital, Aarhus, Central Region Denmark
  - Odense University Hospital, Odense, Region Syddanmark
- Rikshospitalet, Oslo Universitetssykehus, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wareham NE, Mocroft A, Sengelov H, Da Cunha-Bang C, Gustafsson F, Heilmann C, Iversen M, Kirkby NS, Rasmussen A, Sorensen SS, Lundgren JD; MATCH in PERSIMUNE study group. The value of EBV DNA in early detection of post-transplant lymphoproliferative disorders among solid organ and hematopoietic stem cell transplant recipients. J Cancer Res Clin Oncol. 2018 Aug;144(8):1569-1580. doi: 10.1007/s00432-018-2674-9. Epub 2018 May 26. PMID 29804164
- [Background] Allen UD, Preiksaitis JK; AST Infectious Diseases Community of Practice. Post-transplant lymphoproliferative disorders, Epstein-Barr virus infection, and disease in solid organ transplantation: Guidelines from the American Society of Transplantation Infectious Diseases Community of Practice. Clin Transplant. 2019 Sep;33(9):e13652. doi: 10.1111/ctr.13652. Epub 2019 Jul 23. PMID 31230381
- [Result] San-Juan R, Manuel O, Hirsch HH, Fernandez-Ruiz M, Lopez-Medrano F, Comoli P, Caillard S, Grossi P, Aguado JM; ESGICH PTLD Survey Study Group,; European Study Group of Infections in Compromised Hosts (ESGICH) from the European Society of Microbiology and Infectious Diseases (ESCMID). Current preventive strategies and management of Epstein-Barr virus-related post-transplant lymphoproliferative disease in solid organ transplantation in Europe. Results of the ESGICH Questionnaire-based Cross-sectional Survey. Clin Microbiol Infect. 2015 Jun;21(6):604.e1-9. doi: 10.1016/j.cmi.2015.02.002. Epub 2015 Feb 14. PMID 25686696